CLINICAL TRIAL: NCT01864733
Title: Multimodal Approach of Undernutrition in Chronic Heart Failure : a Controlled, Randomized Trial
Brief Title: Multimodal Approach of Undernutrition in Chronic Heart Failure
Acronym: NUTRICARD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Durtol clinical center (Unknown); Centre Hospitalier Universitaire de Saint Etienne (Other); University Hospital, Grenoble (Other); University Hospital, Geneva (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CHU-0152; 2012-A00632-41
Record Dates: First submitted 2013-04-09; First posted 2013-05-30 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Heart Failure
Keywords: Chronic heart failure; Undernutrition; Rehabilitation; Physical exercise; Nutrition; n-3 fatty acids; Androgen; Testosterone
MeSH Terms: conditions — Malnutrition; Motor Activity | interventions — Exercise

ARMS (2):
- intervention group (Experimental): 1) The 'intervention' group: 3-month multimodal approach associating exercise rehabilitation, ONS, n-3 PUFAs and androgen substitution:
  * Physical rehabilitation including endurance and resistance exercises two to three times a week.
  * Oral nutritional supplements: Fortimel max® (Nutricia®) (300 ml, 720 kcal, 29 g de proteins), once per day.
  * n-3 polyunsaturated fatty acids : DHA phospholipids (GPL-DHA®), 240 mg/day.
  * Testosterone: Testopatch® 2.4 mg in men and 1.2 mg in women; 2 patches renewed every two days.
  Interventions: Other: Physical rehabilitation (exercise).
- control group (Other): 2) The 'control' group: no multimodal approach but the treatment currently recommended: heart rehabilitation and dietary counseling during 3 months.
  Interventions: Other: Physical rehabilitation (exercise).

INTERVENTIONS:
Other: Physical rehabilitation (exercise).

SUMMARY:
The treatment of chronic heart failure (CHF) is a key challenge in public health. Despite medical advances, 1-year mortality of NYHA III-IV CHF is 28%. Undernutrition is an independent risk factor for mortality and complications. Up-to-date, interventional studies involving nutrition are scarce in CHF. Academic societies are recommending the use of oral nutritional supplements (ONS) in case of weight loss, without defining the modalities. ONS could improve nutritional status in undernourished CHF patients, but solely administered, have a limited impact on undernutrition, physical performance and prognosis. A multimodal approach integrating physical exercise, nutritional intakes, polyunsaturated n-3 fatty acids (n-3 PUFA), and anabolizing hormones, has to be privileged. A recent trial has shown the clinical benefits of such an approach in patients with chronic respiratory insufficiency (CRI), who have similar nutritional and muscular characteristics.

Exercise rehabilitation is well validated in CHF patients, but has never been validated in case of undernutrition. Exercise rehabilitation allows improving exercise capacity, quality of life and cardiovascular outcomes including mortality.

N-3 PUFA supplementation improves muscle strength and endurance in CRI patients. n-3 PUFA supplementation decreases by 30% cardiovascular mortality of CHF patients. n-3 PUFA could be useful for CHF patients rehabilitation.

Androgenopenia is a prognostic factor in CHF. Androgen substitution improves significantly muscle strength, walking endurance and quality of life. In the context of a multimodal approach, Androgen substitution together with exercise rehabilitation and ONS could have a beneficial effect on muscle mass, strength and endurance of CHF patients, as already described in CRI, elderly and HIV patients.

The study hypotheses that a 3-month multimodal approach associating exercise rehabilitation, androgen substitution, n-3 PUFAs and ONS improves exercise capacity of undernourished CHF patients.

DETAILED DESCRIPTION:
Study aims :

Main study aim :

To evaluate the impact of a 3-month multimodal approach associating exercise rehabilitation, androgen substitution, n-3 PUFAs and ONS on exercise capacity of undernourished CHF patients.

Secondary study aims :

To Evaluate the impact of the 3-month multimodal approach on :

heart function muscle strength exercise endurance body composition and nutritional status quality of life drugs compliance number of hospital stays during one year 1-year survival.

Experimental protocol

Undernourished CHF patients will be randomized into two groups:

1) The 'intervention' group: 3-month multimodal approach associating exercise rehabilitation, ONS, n-3 PUFAs and androgen substitution. 2) The 'control' group: no multimodal approach but the treatment currently recommended: heart rehabilitation and dietary counseling during 3 months.

Both groups will receive by the oral route for 3 months:

vitamin D : 100 000UI/month if plasma 25-OH vitamin D <30 ng/l, ubiquinone : 250 mg/jour in all patients. Both groups will benefit of dietary counseling. A monthly follow-up of compliance will be performed during the 3- month treatment period.

The overall follow-up period will be 15 months, including the 3-month treatment period.

Considering a recruitment period of 18 months and a 15-month follow up, the total study duration will be 33 months.

Primary endpoint: measurement of VO2 at the ventilatory level.

The study hypothesis is to demonstrate in a population of malnourished CHF patients a 10% difference (with a 15% standard error) of the level of VO2 variation between the two groups, measured during the maximal cycle exercise capacity test coupled with respiratory exchanges. VO2 will be measured by the same operators, at baseline and after the 3-month multimodal approach.

Number of subjects to be included :

50 patients per group are needed to demonstrate a 10% difference (with a 15% standard error) if 1st and 2nd error risks respectively fixed at 5% (bilateral) and 10%. Considering the potential studies dropouts, 120 patients will be included.

Inclusion criteria :

Stable patients with CHF, defined by the absence of acute episodes since 2 months, and absence of exercise rehabilitation in the two last months NYHA III Heart failure VO2 peak < 18 ml/kg/min Left ventricle ejection fraction ≤ 40% Age ≥ 18 years, informed, having given their consent Absence of acute disease

Undernutrition, defined by :

Involuntary weight loss ≥5% during the 12 last months, without any increase of diuretics doses or body mass index <20 or fat-free mass index assessed by BIA <18 in men, and <15 in women.

Exclusion criteria :

Heart failure related to pulmonary hypertension Heart failure treatable by surgery or angioplasty Patients eligible to ventricular resynchronisation Instable heart failure Patients waiting for transplantation On-going imunosuppressant or corticosteroids Disease affecting 6-month survival (end-stage cancer, or chronic disease,…) Positive VIH or hepatitis C serology Liver failure Respiratory insufficiency End-stage (stage 5) renal failure (creatinine clearance ≤15ml/kg/min) Acute disease Previous history of hormonal cancer (breast, prostate) Suspected or proved hormonal cancer (breast, prostate) Hypersensibility to testosterone or components of testosterone patch Liver tumor or previous history of liver tumor Unability or contra-indication to rehabilitation program (defined by the French society of Cardiology including contra-indication to physical exercise) Orthopedical limitations to exercise Type 2 diabetes requiring insulin since less than 3 months Patients having not giving their consent.

Statistical analysis STATA V10 (Stata Corp) will be used. The analysis will be performed by intention-to-treat, and, secondly per-protocol. All statistical tests (except for intermediary analysis) will be performed considering a 5% α error risk.

Continuous variables will be presented as mean and standard deviation if normal distribution (Shapiro-Wilk test), and as median, quartiles and extremes, if not. Qualitative variables will be expressed as n (%).

Comparisons between groups will be (1) systematic without any adjustment, and (2) with adjustment on factors not equally distributed between groups despite randomization.

Main endpoint, i.e. ventilatory peak VO2, wil be compared between randomization groups by Student or Kruskal-Wallis tests. Variances equality will be tested with the Fisher-Snedecor test.

In case of adjustment on factors (stratification and treatments), a linear regression model will be performed in the context of a secondary analysis.

Secondary endpoints will be compared according to the same tests and by Chi2 test or exact Fisher test for qualitative parameters.

To measure the variation through time of the different collected parameters, a longitudinal data analysis with ANOVA for repeated data, or Friedman test, followed by a post-hoc test and by mixt models allowing to study inter- or intra-patient variabilities.

Intra-group comparisons will be performed with paired-t Student or Wilcoxon tests for quantitative parameters and Stuart-Maxwell test for qualitative parameters.

12-month survival analysis will be performed according to: univariate analysis: comparison of survival curves with Kaplan-Meier method by log-rank test multivariate analysis with Cox model.

Multivariate analysis models of quality of life (e.g. SF36) will consider the group effect and the patient's demographical/clinical data. To keep a 5% risk for every analysed area, a procedure of 1st species risk correction will be done to calculate the level of significancy of each test.

The rate of expected missing data of the main endpoint was estimated to 20%. A sensitivity analysis of these data will be performed to evaluate its statistical nature: MAR or MCAR and, if necessary it will be decided to use the most appropriate method.

ELIGIBILITY:
Inclusion Criteria:

* Stable patients with CHF, defined by the absence of acute episodes since 2 months, and absence of exercise rehabilitation in the two last months
* NYHA III Heart failure
* VO2 peak < 18 ml/kg/min
* Left ventricle ejection fraction ≤ 40%
* Age ≥ 18 years, informed, having given their consent
* Absence of acute disease
* Undernutrition, defined by :

  * Involuntary weight loss ≥5% during the 12 last months, without any increase of diuretics doses
  * or body mass index <20
  * or fat-free mass index assessed by BIA <18 in men, and <15 in women.

Exclusion Criteria:

* Heart failure related to pulmonary hypertension
* Heart failure treatable by surgery or angioplasty
* Patients eligible to ventricular resynchronisation
* Instable heart failure
* Patients waiting for transplantation
* On-going imunosuppressant or corticosteroids
* Disease affecting 6-month survival (end-stage cancer, or chronic disease,…)
* Positive VIH or hepatitis C serology
* Liver failure
* Respiratory insufficiency
* End-stage (stage 5) renal failure (creatinine clearance ≤15ml/kg/min)
* Acute disease
* Previous history of hormonal cancer (breast, prostate)
* Suspected or proved hormonal cancer (breast, prostate)
* Hypersensibility to testosterone or components of testosterone patch
* Liver tumor or previous history of liver tumor
* Unability or contra-indication to rehabilitation program (defined by the French society of Cardiology including contra-indication to physical exercise)
* Orthopedical limitations to exercise
* Type 2 diabetes requiring insulin since less than 3 months
* Patients having not giving their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
ventilatory workload VO2 | 3 months

SECONDARY OUTCOMES:
Heart function (to measure left ventricle fraction) | at 3 months
Heart function (clinical exam) | at 6 months
Heart function (plasma NT pro-Brain Natriuretic Peptide) | at 3 months
Plasma NT pro-Brain Natriuretic Peptide (Nt ProBNP) | at 3 months and at 6 months
Maximal cycle exercise capacity test coupled with respiratory exchanges: VO2 peak, peak workload on bicycle, endurance time between peak and ventilatory workload | at 3 months
Quadriceps strength | at 3 months
6-min walking test | at 3 months
Nutritional status (weight, height, body mass index) | before intervention and at 3 months and 6 months
Quality of life with specific questionnaires | before intervention and at 3 months and 6 months
Hospital stays (number of days) | at 12 months and at 15 months
Body composition (weight, height, body mass index) | at month 3 and month 6

CONTACTS AND LOCATIONS:
Overall Officials: Ronan THIBAULT, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France